CLINICAL TRIAL: NCT06868342
Title: Determination of Feasibility of Reversible Conduction Block Generated Using Peripheral Nerve Stimulator in Treatment of Focal Spasticity and the Stimulation Parameters for the Same.
Brief Title: Nerve Root Block in Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walton Centre NHS Foundation Trust (Other)
Collaborators: Nevro Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RG420-21
Record Dates: First submitted 2025-03-07; First posted 2025-03-10 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Spasticity; Spasticity in Participants With Multiple Sclerosis; Spasticity Post Stroke; Spasticity Related to Any Cause Except Cerebral Palsy
Keywords: Spasticity; High-Frequency Stimulation; Electrical Nerve Block; Conduction Block
MeSH Terms: conditions — Muscle Spasticity; Heart Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nerve block (Experimental): The group of participants undergoing tibial neurectomy for focal spasticity to whom the high frequency nerve conduction block shall be applied.
  Interventions: Procedure: High-frequency nerve conduction block

INTERVENTIONS:
Procedure: High-frequency nerve conduction block — A high-frequency nerve conduction block applied to a muscular branch of the tibial nerve and assessed by intraoperative EMG, performed before the nerve is cut as a part of a standard tibial neurectomy for focal spasticity.
  Other Names: HFNB

SUMMARY:
In this work the investigators propose to briefly apply kilohertz frequency alternating current via PNS device placed next to the isolated nerve in 4 patients undergoing peripheral neurectomy, just before cutting the nerve. The intervention shall be performed utilizing EMG monitoring and mapping. After the muscular branches of the tibial nerve are exposed, proximal stimulation (1Hz) shall be applied to a selected branch with a bipolar electrode to produce muscle contractions. A high frequency (10kHz) blocking current shall be applied by placing a PNS electrode distally to the bipolar electrode and the EMG shall be recorded. The PNS electrode shall be removed from surgical field and further proximal stimulation done to confirm reversal of block (return to baseline) on the EMG. Then the nerve will be severed as a part of standard tibial neurectomy, and further proximal and distal stimulation shall be performed. The results will be compared to see if high frequency conduction block can physiologically mimic peripheral neurectomy; and obtain parameters of stimulation required for that.

DETAILED DESCRIPTION:
Dysregulated neural activity is responsible for many ailments- focal spasticity after stroke or spinal cord injury, reflex incontinence, overactive bladder, etc. Current treatment options for such pathologies are suboptimal and include ablative procedures like neurectomy. Neurectomy inadvertently leads to loss of function. Modulated electrical conduction block can help control this activity without causing additional loss of function and thus has immense potential in treatment of these conditions.

Animal experiments have suggested that such a block is feasible. While safety ranges for delivery of current to human peripheral nerves are known and stimulation parameters for activation of nerves well established, further data is needed to assess the parameters for clinically useful conduction block. Currently such data studies are being conducted to block pain from neuroma after amputation and to block vagal nerve for obesity.

Peripheral Neurectomy is a procedure used for treating focal spasticity when less invasive options have been unsuccessful. The procedure is performed under full Neurophysiology monitoring. Intra-operatively, the nerve is exposed and motor activity from this is recorded spontaneously and with direct bipolar stimulation with help of EMG electrodes placed in the territory of the nerve. A tetanic response obtained upon such stimulation indicates spasticity. The nerve is cut, and further testing done by stimulating proximal and distal to the cut. Lack of tetanic response after proximal stimulation indicates adequacy of procedure.

In this work the investigators propose to briefly apply kilohertz frequency alternating current via PNS device placed next to the isolated nerve in 4 patients undergoing peripheral neurectomy, just before cutting the nerve. The intervention shall be performed utilizing EMG monitoring and mapping. After the muscular branches of the tibial nerve are exposed, proximal stimulation (1Hz) shall be applied to a selected branch with a bipolar electrode to produce muscle contractions. A high frequency (10kHz) blocking current shall be applied by placing a PNS electrode distally to the bipolar electrode and the EMG shall be recorded. The PNS electrode shall be removed from surgical field and further proximal stimulation done to confirm reversal of block (return to baseline) on the EMG. Then the nerve will be severed as a part of standard tibial neurectomy, and further proximal and distal stimulation shall be performed. The results will be compared to see if high frequency conduction block can physiologically mimic peripheral neurectomy; and obtain parameters of stimulation required for that.

This will be a proof of concept work assessing feasibility of conduction block for focal spasticity. If successful, further pilot study shall be done to assess efficacy.

Apart from brief application of high frequency stimulation, the rest of the procedure will be standard.

The stimulation will be within parameters approved by FDA and CE marking. As the nerve will then be cut anyway, there is no additional risk of harm to the nerve or the patient.

This study will adhere to the principles outlined in the UK Policy Framework for Health and Social Care Research (v3.2 10th October 2017). It will be conducted in compliance with the protocol, the EU General Data Protection Regulation 2016 and Data Protection Act 2018, and other regulatory requirements as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above selected for peripheral neurectomy for focal spasticity
* Functioning LMN pathway determined by EMG

Exclusion Criteria:

* Age <18yr
* Myopathy and other LMN disorders
* Impaired LMN pathway determined by EMG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
EMG - Nerve conduction block | Intraoperative.
  Following the application of the high-frequency current to the distal part of the nerve, the stimulated EMG shall show the decrease in amplitude [uV], compared to baseline EMG.
EMG - The reversibility of nerve conduction block | Intraoperative.
  After stopping the high-frequency stimulation, the stimulated EMG amplitudes shall return to baseline [uV].
EMG - Comparative analysis of the effects of nerve block vs. neurectomy. | Intraoperative
  After the nerve block is reversed, a standard tibial neurectomy shall be performed. Stimulated EMG amplitudes [uV] shall be compared to those recorded at the time of nerve block [uV].

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Marshall, PhD, Study Chair — Walton Centre NHS Foundation Trust
Locations (1):
- The Walton Centre NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The data generated during the study comprises of EMG recordings stored on the password protected computers within the Trust. The anonymised EMG data for each participant shall be disseminated as a part of a publication.

REFERENCES:
- [Background] Sitthinamsuwan B, Chanvanitkulchai K, Phonwijit L, Ploypetch T, Kumthornthip W, Nunta-Aree S. Utilization of intraoperative electromyography for selecting targeted fascicles and determining the degree of fascicular resection in selective tibial neurotomy for ankle spasticity. Acta Neurochir (Wien). 2013 Jun;155(6):1143-9. doi: 10.1007/s00701-013-1686-0. Epub 2013 Apr 7. PMID 23563747
- [Background] Deer TR, Naidu R, Strand N, Sparks D, Abd-Elsayed A, Kalia H, Hah JM, Mehta P, Sayed D, Gulati A. A review of the bioelectronic implications of stimulation of the peripheral nervous system for chronic pain conditions. Bioelectron Med. 2020 Apr 24;6:9. doi: 10.1186/s42234-020-00045-5. eCollection 2020. PMID 32346553
- [Background] Mikalef P, Power D. The role of neurectomy in the management of spasticity of the upper limb. EFORT Open Rev. 2017 Nov 27;2(11):469-473. doi: 10.1302/2058-5241.2.160074. eCollection 2017 Nov. PMID 29218232
- [Background] Yong LY, Wong CHL, Gaston M, Lam WL. The Role of Selective Peripheral Neurectomy in the Treatment of Upper Limb Spasticity. J Hand Surg Asian Pac Vol. 2018 Jun;23(2):181-191. doi: 10.1142/S2424835518500182. PMID 29734901
- [Background] Van Buyten JP, Al-Kaisy A, Smet I, Palmisani S, Smith T. High-frequency spinal cord stimulation for the treatment of chronic back pain patients: results of a prospective multicenter European clinical study. Neuromodulation. 2013 Jan-Feb;16(1):59-65; discussion 65-6. doi: 10.1111/ner.12006. Epub 2012 Nov 30. PMID 23199157
- [Background] Camilleri M, Toouli J, Herrera MF, Kow L, Pantoja JP, Billington CJ, Tweden KS, Wilson RR, Moody FG. Selection of electrical algorithms to treat obesity with intermittent vagal block using an implantable medical device. Surg Obes Relat Dis. 2009 Mar-Apr;5(2):224-9; discussion 229-30. doi: 10.1016/j.soard.2008.09.006. Epub 2008 Sep 12. PMID 18996767
- [Background] Soin A. Long-term human testing of high-frequency nerve block for amputation pain. Paper presented at: 16th Annual Meeting North American Neuromodulation Society; December 6 to 9, 2012; Las Vegas, NV, USA.
- [Background] Perruchoud C, Eldabe S, Batterham AM, Madzinga G, Brookes M, Durrer A, Rosato M, Bovet N, West S, Bovy M, Rutschmann B, Gulve A, Garner F, Buchser E. Analgesic efficacy of high-frequency spinal cord stimulation: a randomized double-blind placebo-controlled study. Neuromodulation. 2013 Jul-Aug;16(4):363-9; discussion 369. doi: 10.1111/ner.12027. Epub 2013 Feb 20. PMID 23425338
- [Background] Bhadra N, Vrabec TL, Bhadra N, Kilgore KL. Reversible conduction block in peripheral nerve using electrical waveforms. Bioelectron Med (Lond). 2018 Jan;1(1):39-54. doi: 10.2217/bem-2017-0004. Epub 2017 Dec 14. PMID 29480897
- [Background] Kilgore KL, Bhadra N. Nerve conduction block utilising high-frequency alternating current. Med Biol Eng Comput. 2004 May;42(3):394-406. doi: 10.1007/BF02344716. PMID 15191086